CLINICAL TRIAL: NCT01592123
Title: Evaluation of Benefits of Nasal Septal Surgery on Subjective Sleep Quality, Daytime and Dream Anxiety
Brief Title: Effects of Nasal Septal Surgery on Sleep Quality, Daytime and Dream Anxiety
Status: Completed | Type: Observational
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Gulec, M.D., Psych., Assist. Prof., M.D., Psych., Assist. Prof., Ataturk Training and Research Hospital
Other Study IDs: MG-ATA-001
Record Dates: First submitted 2012-04-30; First posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Nasal Septal Deviation
Keywords: anxiety; septal surgery; septum deviation; sleep
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The participants with septal deviation
  Interventions: Procedure: The active anterior rhinomanometry; Behavioral: The Pittsburgh Sleep Quality Index (PSQI); Behavioral: The Beck Anxiety Inventory (BAI); Behavioral: The Van Dream Anxiety Scale (VDAS)

INTERVENTIONS:
Procedure: The active anterior rhinomanometry — In this method, the airflow through 1 nasal cavity and the pressure gradient across this nasal cavity are measured simultaneously at each breath as recommended by the committee report on the standardization of rhinomanometry. All measurements were performed under the same standard conditions. Herein, all presented airflow values are the sum of inspiratory airflow of the right and left sides of the nose at 150 pascals (Pa). And, total nasal airflow (cm3/s) and airway resistance (Pa/cm3/s) values were used for statistical analyses.
  Other Names: Rhino 4000M (Homoth, Hamburg, Germany)
Behavioral: The Pittsburgh Sleep Quality Index (PSQI) — PSQI was developed to measure sleep quality during the previous month and to discriminate between good and poor sleepers. The self-administered scale contains 15 multiple-choice items that inquire about frequency of sleep disturbances and subjective sleep quality and 4 write-in items that inquire about typical bedtime, wake-up time, sleep latency, and sleep duration. Each component score ranges from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range of 0-21). A PSQI global score >5 is considered to be suggestive of significant sleep disturbance.
  Other Names: The Pittsburgh Sleep Quality Index (Buysse et al., 1989)
Behavioral: The Beck Anxiety Inventory (BAI) — The BAI is a 21-item self-report questionnaire that lists symptoms of anxiety. The respondent is asked to rate how much each symptom has bothered him/her in the past week. The symptoms are rated on a four-point scale, ranging from ''not at all'' (0) to ''severely'' (3). The instrument has excellent internal consistency and high test-retest reliability. The BAI has been widely used to measure severity of anxiety by self-report.
  Other Names: The Beck Anxiety Inventory (Beck et al., 1988)
Behavioral: The Van Dream Anxiety Scale (VDAS) — The VDAS provides the assessment of nightmare frequency and dream anxiety caused by frightening dreams during the preceding month. There are 17 self-rated questions in the scale. Twelve questions (1-4, 6, 11-17) that are tabulated in the scoring are weighted equally on a 0-4 scale. Question 5 is related to autonomic hyperactivity and consists of 12 symptoms. Each of 12 symptoms is also weighted on a 0-4 scale. Thirteen question scores are summed to yield a global VDAS score, which has a range of 0-42.
  Other Names: The Van Dream Anxiety Scale (Agargun et al., 1999)

SUMMARY:
The aim of this report was to assess the frequency of poor sleep quality, daytime and dream anxiety and their response to subsequent surgical treatment for a representative group patients with nasal septum deviation.

DETAILED DESCRIPTION:
Prior to the surgery, nasal airflows and airway resistances were measured employing rhinomanometry and they were also asked to fill in the Pittsburgh Sleep Quality Index (PSQI), the Beck Anxiety Inventory (BAI), and the Van Dream Anxiety Scale (VDAS). And, a postoperative assessment for the same parameters was made at two months from the day of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* All participants, 18 to 65 years of age, had septal deviation consistent with the presenting symptoms which last at least three months and persist after a three months trial of medical management, including topical nasal steroids, topical or oral decongestants, or an oral antihistamine/decongestant combination.

Exclusion Criteria:

Patients were excluded from the study if they had nasal septal surgery performed for other reasons, such as

* an access to nasal and sinus tumors,
* pituitary surgery and as part of treatment for sleep apnea or with concurrent sinus surgery;
* had rhinoplasty prior to submucous resection;
* had acute nasal trauma;
* had adenoid hypertrophy;
* had uncontrolled asthma/nasal allergy;
* had diagnosed or suspected (snoring with/without other symptoms, such as apneas referred by someone and/or somnolence) OSA;
* had obesity (BMI ≥ 30.0 kg/m2);
* had an unstable physical disorder;
* had a current or lifetime history of any functional or organic mental disorder;
* had a history of seizures;
* had a neurological disorder that significantly affects central nervous system functions;
* had met criteria for substance abuse or dependence in the previous 12 months, including nicotine dependence;
* were taking medications that may cause or exacerbate sleep problems, daytime and dream anxiety; had clinical or laboratory evidence of hypothyroidism without adequate and stable replacement therapy;
* had a history of antidepressant or sedative-hypnotic medications for any current or past complaint;
* were pregnant or breastfeeding; or
* were women not using effective contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Otorhinolaryngology outpatient clinic
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-10; Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The amelioration of subjective sleep quality with nasal septal surgery. | A postoperative assessment for the aforementioned parameter was made at two months from the day of the surgery.
  The Pittsburgh Sleep Quality Index (PSQI) was used for the evaluations.
The amelioration of daytime anxiety with nasal septal surgery. | A postoperative assessment for the aforementioned parameter was made at two months from the day of the surgery.
  The Beck Anxiety Inventory (BAI) was used for the evaluations.
The amelioration of dream anxiety with nasal septal surgery. | A postoperative assessment for the aforementioned parameter was made at two months from the day of the surgery.
  The Van Dream Anxiety Scale (VDAS) was used for the evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Gulec, investigator, Principal Investigator — Ataturk University, Faculty of Medicine, Department of Psychiatry
Locations (1):
- Ataturk University, Yakutiye Research Hospital, Erzurum, Yakutiye, Turkey (Türkiye)

REFERENCES:
- [Background] Baumann I. Quality of life before and after septoplasty and rhinoplasty. GMS Curr Top Otorhinolaryngol Head Neck Surg. 2010;9:Doc06. doi: 10.3205/cto000070. Epub 2011 Apr 27. PMID 22073110
- [Background] Moore M, Eccles R. Objective evidence for the efficacy of surgical management of the deviated septum as a treatment for chronic nasal obstruction: a systematic review. Clin Otolaryngol. 2011 Apr;36(2):106-13. doi: 10.1111/j.1749-4486.2011.02279.x. PMID 21332671